CLINICAL TRIAL: NCT06070233
Title: A Randomized, Sham Controlled Trial of Dorsal Root Rhizotomy Stereotactic Radiosurgery Versus Standard of Care for Spasticity Associated With Stroke, Spinal Cord Injury & Cerebral Palsy
Brief Title: Radiosurgery Treatment for Spasticity Associated With Stroke, SCI & Cerebral Palsy
Acronym: SPASM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ohio State University (Other)
Collaborators: Varian Medical Systems (Industry)
Responsible Party: Principal Investigator, Joshua Palmer, Professor, Radiation Oncology, Ohio State University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 2022H0425
Record Dates: First submitted 2023-09-30; First posted 2023-10-06 (Actual); Last update posted 2025-12-19 (Actual); Status verified 2025-12

CONDITIONS: Spasticity as Sequela of Stroke; Spastic Cerebral Palsy; Spasticity, Muscle
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity | interventions — Radiosurgery; Spermine Synthase; salicylhydroxamic acid

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Sham Treatment (Sham Comparator): No intervention but can crossover after 6 months
  Interventions: Other: Sham
- SRS Treatment (Active Comparator)
  Interventions: Radiation: stereotactic radiosurgery (SRS) dorsal root rhizotomy radiomodulation

INTERVENTIONS:
Radiation: stereotactic radiosurgery (SRS) dorsal root rhizotomy radiomodulation — Patients will be simulated in the supine position in an immobilization apparatus deemed by the treating physician to be appropriate for the patient being able to comfortably maintain position for the duration of treatment. All patients will be simulated and treated using free breathing. Prescription dose is 50 Gy delivered in a single fraction to the target volume, prescribed to whatever isodose line produces optimal falloff (but not less than a 50% isodose line; dmax <100Gy) .
  All radiosurgery treatment will utilize the Varian Edge, Varian TrueBeam STx, or CyberKnife system
  Arms: SRS Treatment
Other: Sham — Patients will be simulated in the supine position in an immobilization apparatus deemed by the treating physician to be appropriate for the patient being able to comfortably maintain position for the duration of treatment. All patients will be simulated and treated using free breathing.
  Arms: Sham Treatment

SUMMARY:
A scientific study is being done to test a special treatment for people who have spasticity or tight muscles. This treatment is called "stereotactic radiosurgery dorsal rhizotomy." It uses very accurate beams of radiation to target certain nerves in the back to help loosen up the muscles. In this study, people are put into two groups by chance: one group gets the real treatment, and the other group gets a "fake" treatment that doesn't do anything. This fake treatment is called a "sham." Doing this helps make sure the study is fair and the results are true. After the people in the study get their treatment, the researchers will watch and see how they do. They will check if their muscles are less stiff and if they have any side effects. By looking at the results from both groups, the researchers can find out if the special treatment really helps people with spasticity. Patients who got the "fake" treatment will be eligible to receive the "real" treatment after 6 months.

ELIGIBILITY:
Inclusion Criteria:

* Chronic spasticity refractory to medical management or in a patient who cannot receive appropriate medical management mediated by one or more spinal nerve roots
* Age > 16 (if under 18, patients parents must sign consent).

Exclusion Criteria:

* Inability to lie supine for simulation & treatment
* Inability to visualize the target nerve on either CT or MRI imaging
* Patients with confirmed pregnancy (all women of child-bearing age with intact uterus & ovaries will be required to undergo a pregnancy test prior to simulation)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22 (Estimated)
Dates: Start 2023-10-12 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Modified Ashworth Scale | 6 months post treatment
  Change in the 6-month post-treatment Modified Ashworth Scale (MAS) measure of spasticity, which ranges from 0 (no symptoms) to 4 (worst symptoms)

SECONDARY OUTCOMES:
Change in spasticity-related quality of life (SQoL-6D) | 2 years post treatment
  Change in spasticity-related quality of life 6-dimensions instrument (SQoL-6D) over two years post-treatment, where the scale ranges from 0 (worst quality of life) to 100 (best quality of life)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Palmer, MD, Principal Investigator — Ohio State University
Locations (2):
- United States (2):
  - Renaissance Institute of Precision Oncology & Radiosurgery, Winter Park, Florida
  - Ohio State University Wexner Medical Center, Columbus, Ohio

DOCUMENTS (1):
  • Informed Consent Form (2023-09-22): https://cdn.clinicaltrials.gov/large-docs/33/NCT06070233/ICF_000.pdf